CLINICAL TRIAL: NCT04928144
Title: An Intra-subject Dose Escalation Phase 1 Study to Determine the Safety and Tolerability of SHJ002 Sterile Ophthalmic Solution in Pediatric Subjects
Brief Title: Phase 1 Study of SHJ002 Sterile Ophthalmic Solution in Pediatric Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunhawk Vision Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SHJ002-CS201
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Myopia
Keywords: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Single-center, Open-label, first-in-human dose-escalation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 0.025% SHJ002 (Experimental): 0.025% SHJ002 Sterile Ophthalmic Solution
  Interventions: Drug: SHJ - Low concentration
- 0.080% SHJ002 (Experimental): 0.080% SHJ002 Sterile Ophthalmic Solution
  Interventions: Drug: SHJ - Mid concentration
- 0.25% SHJ002 (Experimental): 0.25% SHJ002 Sterile Ophthalmic Solution
  Interventions: Drug: SHJ - High concentration
- SHJ002 - Maximum tolerated concentration (Experimental): Maximum tolerated concentration of SHJ002
  Interventions: Drug: SHJ - Maximum tolerated

INTERVENTIONS:
Drug: SHJ - Low concentration — Topical ophthalmic
  Arms: 0.025% SHJ002
Drug: SHJ - Mid concentration — Topical ophthalmic
  Arms: 0.080% SHJ002
Drug: SHJ - High concentration — Topical ophthalmic
  Arms: 0.25% SHJ002
Drug: SHJ - Maximum tolerated — SHJ - Maximum tolerated
  Arms: SHJ002 - Maximum tolerated concentration

SUMMARY:
This is a single-center, open-label, first-in-human dose-escalation study of SHJ002 Ophthalmic Solution in children. (Part 1) Three (3) subjects will receive each concentration of SHJ002 for 3 days in an escalation design in one eye. (Part 2) A Group of 9 additional children will receive the highest tolerated concentration for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Non-cycloplegic sphere from +1.50 to -4.75 Diopters in one or both eyes.
* A minor able to complete all study assessments and comply with the protocol and has a parent or caregiver willing and able to follow study instructions, comply with the protocol and attend study visits with the subject as required, in the opinion of the Investigator.
* Literate and able to orally communicate.

Exclusion Criteria:

* Non-cycloplegic sphere worse than -4.75 Diopters
* Axial length > 26 mm
* Hyperopia worse than +1.50 Diopters
* Anisometropia (difference of myopic power >2.00 D).
* Astigmatism > 1.5 D.
* Intraocular pressure > 21 mm Hg or < 6 mm Hg.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-09-17 (Actual)

PRIMARY OUTCOMES:
Change from baseline in best corrected visual acuity | 3 days (Part 1) and 28 days (Part 2)
  Change from baseline in best corrected visual acuity
Incidence of Adverse Events | 3 days (Part 1) and 28 days (Part 2)
  Incidence of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Suh-Hang H. Juo, MD, Ph.D., Study Director — Sunhawk Vision Biotech, Inc.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen JL, Lai WY, Lin RT, Juo SH, Liang CL. Safety and Tolerability of Anti-microRNA-328 Ophthalmic Solution, SHJ002, in Pediatric Subjects: First-in-Human Clinical Study. Clin Ther. 2024 Oct;46(10):768-772. doi: 10.1016/j.clinthera.2024.08.015. Epub 2024 Sep 7. PMID 39244490